CLINICAL TRIAL: NCT00476073
Title: Efficacy and Safety of Flutiform® pMDI in Adult Patients With Mild to Moderate-severe Reversible Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: FLT3501
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Asthma Bronchiale
MeSH Terms: interventions — fluticasone-formoterol; Formoterol Fumarate; Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: FLUTIFORM® (Formoterol fumarate / Fluticasone propionate)

SUMMARY:
Open, parallel group design. The study has a screening phase and a 12 week treatment phase. Subjects will be randomised to treatment in a 1:1 ration.

DETAILED DESCRIPTION:
This is a study involving a 12 week treatment phase. During the treatment phase subjects receive FLUTIFORM® or Sertetide®. Efficacy will be assessed by lung function tests and asthma symptoms, sleep disturbance. Safety will be assessed by adverse events, vital signs, lab tests and ECGs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients at least 18 years or older (females less than one year post-menopausal must have a negative serum or urine pregnancy test recorded within 72 hours prior to the first dose of study medication, be non-lactating, and willing to use adequate and highly effective methods of contraception throughout the study. A highly effective method of birth control is defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as sterilization, implants, injectables, combined oral contraceptives, some IUDs (Intrauterine Device, hormonal), sexual abstinence or vasectomised partner).
* Known history of mild to moderate-severe reversible asthma for > 6 months prior to the screening visit.
* Demonstrate a FEV1 of >40% to <80% for predicted normal values (EGKS normal values, 1983) during the screening phase following appropriate withholding of asthma medications (if applicable).

  * No beta agonist use on day of screening.
  * No use of combination asthma therapy on day of screening.
  * Inhaled corticosteroids are allowed on day of screening.
* Documented reversibility of > 15% in FEV1 in the screening phase.
* Demonstrate satisfactory technique in the use of the pressurized MDI.
* Willing and able to enter information in the electronic diary and attend all study visits.
* Willing and able to substitute study medication for their pre study prescribed asthma medication for the duration of the study.
* Written informed consent obtained.

Exclusion Criteria:

* Life-threatening asthma within the past year. This category includes those patients with a history of near-fatal asthma, a hospitalization or an emergency visit for asthma or prior intubation for asthma.
* History of systemic (injectable) corticosteroid medication within 1 month before the Screening Visit.
* History of omalizumab use within the past 6 months.
* History of leukotriene receptor antagonist use, e.g. montelukast, within the past week.
* Current evidence or history of any clinically significant disease or abnormality including uncontrolled coronary artery disease, congestive heart failure, myocardial infarction, or cardiac dysrhythmia. 'Clinically significant' is defined as any disease that, in the opinion of the Investigator, would put the patient at risk through study participation, or which would affect the outcome of the study.
* An upper or lower respiratory infection within 4 weeks prior to the Screening Visit.
* Significant, non-reversible, active pulmonary disease (e.g., chronic obstructive pulmonary disease (COPD), cystic fibrosis, bronchiectasis, tuberculosis).
* Known Human Immunodeficiency Virus (HIV)-positive status.
* A smoking history equivalent to "10 pack years" (i.e., at least 1 pack of 20 cigarettes /day for 10 years or 10 packs/day for 1 year, etc)
* Current smoking history within 12 months prior to the Screening Visit.
* Current evidence or history of alcohol and/or substance abuse within 12 months prior to the Screening Visit.
* Patients who have taken beta-blocking agents, tricyclic antidepressants, monoamine oxidase inhibitors, astemizole (Hismanal), quinidine type antiarrhythmics, or potent CYP 3A4 inhibitors such as ketoconazole within the past week.
* Current use of medications that will have an effect on bronchospasm and/or pulmonary function.
* Current evidence or history of hypersensitivity or idiosyncratic reaction to test medications or components.
* Receipt of an investigational drug within 30 days of the Screening Visit (12 weeks if an oral or injectable steroid).
* Current participation in a clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2007-04; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
FEV1, (Forced expiratory volume in the 1st second).

SECONDARY OUTCOMES:
Other lung function tests, AQLQ, Safety Assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Blagden, MD, Principal Investigator
Locations (1):
- Dr Blagden, Chesterfield, United Kingdom

REFERENCES:
- [Derived] Aalbers R, Brusselle G, McIver T, Grothe B, Bodzenta-Lukaszyk A. Onset of bronchodilation with fluticasone/formoterol combination versus fluticasone/salmeterol in an open-label, randomized study. Adv Ther. 2012 Nov;29(11):958-69. doi: 10.1007/s12325-012-0058-0. Epub 2012 Oct 17. PMID 23081745
- [Derived] Bodzenta-Lukaszyk A, Dymek A, McAulay K, Mansikka H. Fluticasone/formoterol combination therapy is as effective as fluticasone/salmeterol in the treatment of asthma, but has a more rapid onset of action: an open-label, randomized study. BMC Pulm Med. 2011 May 23;11:28. doi: 10.1186/1471-2466-11-28. PMID 21605396
- See also: Related Info — https://www.clinicaltrialsregister.eu/ctr-search/search?query=FLT3501
- See also: Results posted on Eu Clinical Trials Register — https://www.clinicaltrialsregister.eu